CLINICAL TRIAL: NCT04426799
Title: Lemon Essential Oil in Reducing Test Anxiety
Brief Title: Effectiveness of Lemon Essential Oil of Aromatherapy in Reducing Test Anxiety in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, ASSISTANT PROFESSOR, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/1
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Nursing Student
Keywords: Lemon Essential Oil; Test Anxiety,; Student; Nurse

STUDY DESIGN:
Intervention Model Description: : A randomized, pre-test-post-test design was carried out to examine the effectiveness of lemon essential oil in reducing test anxiety in first-year students of the Faculty of Medical Sciences of a private university in Istanbul.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): no application
- Experimental group (Experimental): application is done
  Interventions: Other: lemon essential oil

INTERVENTIONS:
Other: lemon essential oil — A randomized, pre-test-post-test design was carried out to examine the effectiveness of lemon essential oil in reducing test anxiety in first-year students of the Faculty of Medical Sciences of a private university in Istanbul
  Arms: Experimental group

SUMMARY:
This study examines the effectiveness of lemon essential oil in reducing test anxiety in first-year nursing students.

DETAILED DESCRIPTION:
While studies on the role of aromatherapy in reducing test anxiety exist, those evaluating the effects of lemon essential oil on test anxiety are extremely limited. In this study, the effect of a different aromatherapy application on reducing test anxiety was tried to be determined by using lemon essential oil. It is envisaged to provide an alternative aromatherapy application to students and educators to reduce test anxiety through the results obtained in the study.

ELIGIBILITY:
Inclusion Criteria:

* No respiratory system diseases (Asthma, Flu etc.)
* no allergy to any smell, no pregnancy status,
* absence of epilepsy discomfort,
* not having a condition that prevents smell, not using any medication that will affect heart rate and blood pressure,

exclusion criteria

* Any respiratory system disease (Asthma, Flu, etc.).
* have a known allergic response to essential oil to be used,
* Lack of smell, use of any medication affecting heart rate and blood pressure,
* to use other complementary medicine practices

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 30 minutes
  The personal information form contained nine questions on age, gender, education level, profession, place of residence, socio-economic status and total GPA (Grade Point Average).
Test Anxiety Scale (TAS) | 30 minutes
  Developed by Bozkurt (2019), the scale evaluates the degree of anxiety students feel before a test on a scale of 0 to 10. A score of 0 indicates no anxiety, while a score of 10 indicates severe anxiety 28
State Test Anxiety Scale | 30 minutes
  Developed by Şahin in 2019, this scale determines students' anxiety levels before a test. It is a 4-point Likert-type scale consisting of three sub-dimensions and 22 items. The cognitive dimension consists of nine items (3, 4, 7, 9, 14, 16, 18, 20, 22), wherein the lowest possible score is nine and the highest score is 36. The psychosocial dimension consists of five items (6, 10, 12, 13, 21), wherein the lowest possible score is 5 and the highest score is 20. The physiological dimension includes eight items (1, 2, 5, 8, 11, 15, 17, 19), wherein the lowest possible score is 8 and the highest score is 32. Possible scores on the scale ranged between 22 and 88

CONTACTS AND LOCATIONS:
Overall Officials: Züfünaz Özer, Principal Investigator — Sabahattin Zaim University
Locations (1):
- Sabahattin Zaim University, Istanbul, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT04426799/Prot_SAP_000.pdf